CLINICAL TRIAL: NCT06882798
Title: A New Clinical Model for the Engagement of Latinx Youth With Suicidal Behavior and Their Families in a Culturally Centered CBT Treatment
Brief Title: A New Clinical Model for the Engagement of Latinx Youth With Suicidal Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STR-1-138-22
Record Dates: First submitted 2025-03-17; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Suicide Ideation; Suicidal Behaviors; Depressive Symptoms
Keywords: Suicidal Ideation; Suicide Attempt; Randomized controlled trial; adolescents; Latinx; Latina; Latino; Hispanic; cognitive behavioral therapy; depressive symptoms; community health workers
MeSH Terms: conditions — Depression; Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCBT-SB (Only) (Active Comparator): A culturally centered CBT treatment protocol called Socio-Cognitive Behavioral Therapy for Suicidal Behavior (SCBT-SB)
  Interventions: Behavioral: Socio-Cognitive Behavioral Therapy for Suicidal Behavior (SCBT-SB)
- New Clinical Model: SCBT-SB + Community Health Worker (Experimental): SCBT-SB treatment with the additional support of a community health worker (CHW)
  Interventions: Behavioral: SCBT-SB + CHW

INTERVENTIONS:
Behavioral: Socio-Cognitive Behavioral Therapy for Suicidal Behavior (SCBT-SB) — SCBT-SB is a manualized psychosocial treatment protocol developed specifically with and for L/H youth with suicidal ideation and behaviors. Clinician, adolescents, and caregivers' manuals are available in both Spanish and English. SCBT-SB protocol's main conceptual framework and strategies are informed by Cognitive Behavioral Therapy concepts, psychoeducation, and adolescent parenting strategies. The intervention involves individual, caregivers, and family sessions. SCBT-SB, while maintaining the basic principles of CBT, was further developed to include developmental (e.g., identity), and cultural elements of L/H families (e.g., family communication, language). The protocol has two main phases. Phase 1, the Crisis Module, includes nine standard core sessions, and Phase 2, which proposes a flexible number of sessions, focused on the delivery of interchangeable coping skills modules and the acquisition of skills that reduce STB.
  Arms: SCBT-SB (Only)
Behavioral: SCBT-SB + CHW — The New Clinical Model consist of one clinician delivering the SCBT-SB and one CHW per each family. The assigned clinician & CHW will meet at the beginning of treatment to discuss their assigned case and will have follow-up meetings as needed and at a minimum, once monthly. CHWs will support family engagement in treatment. CHWs will assess each family's social needs and concerns about treatment. The CHW intervention will 1) Assess social determinants of mental health; 2) Provide referrals and serve as a bridge to other community resources; 3) Provide psychoeducation on mental health and services to decrease stigma; and 4) Follow-up and provide support on recommended actions.
  Arms: New Clinical Model: SCBT-SB + Community Health Worker

SUMMARY:
This study will test a model of providing treatment to Latinx/Hispanic youth, who experience suicidal thoughts and behavior, and their caregivers. An affirmative and culturally relevant treatment will be provided to all youth and half of the families will be assigned to the additional support of a community health worker (CHW). Youth symptoms and family engagement to treatment will be followed for nine months. The potential benefit of adding the CHW intervention will be assessed.

DETAILED DESCRIPTION:
The objective of this proposal is to test a New Clinical Model to engage Latinx/Hispanic (L/H) youth and their caregivers in a culturally centered, evidence-based treatment for suicidal behaviors (SB). The Socio-Cognitive Behavioral Therapy for Suicidal Behavior (SCBT-SB) is an affirmative and culturally relevant treatment with empirical evidence supporting its use for L/H youth with suicidality. The New Clinical Model consists of the addition of community health workers (CHWs) to the SCBT-SB. CHWs are trusted members of their communities who provide education and connection to resources to L/H families in their native language. A community based participatory research approach is proposed and the Socio-Cultural Framework for Health Service Disparities will be the theoretical model used.

ELIGIBILITY:
Inclusion Criteria:

* Latinx, defined as have been born in a Latin country or having at least one biological parent, grandparent or an ancestor that was born in a Latin country
* Severe Suicidal Ideation (SI), defined as one of the following:
* SIQ-JR > 22 or endorsing any critical items (2, 3, 4, 7, 8, 9) with at least "about 1x/month"
* CDI-II > 15 and endorsing "I think about killing myself but would not do it" OR "I think about killing myself."
* PHQ-9 > 10 & endorsing the item "Thoughts that you would be better off dead, or of hurting yourself in some way" with a frequency of "several days" or greater or endorsing the item "Has there been a time in the past month when you have had serious thoughts about ending your life?
* Suicidal crisis within the past 12 months
* Caregivers and adolescents fluent in Spanish or English language and legal guardian willing to participate

Exclusion Criteria:

* Participants will be referred to a different treatment program if their main clinical complaint is any of the following:
* Behavioral (e.g., conduct disorder, or substance use disorder)
* An eating disorder
* Obsessive-compulsive disorder
* A developmental issue (e.g., speech, occupational, families looking for assessments, treatment for autism) or a significant cognitive delay that may require specialized treatment adjustments.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation (SI) | Change from baseline to 6 months and baseline to 9 months.
  Suicidal ideation measured using the Suicide Ideation Questionnaire-Junior (SIQ-JR), a self-report instrument of 15 items that measures severity of suicidal ideation as a continuous variable with established normative, reliability, and validity data for clinical and non-clinical adolescent samples. The minimum score is 0 and the maximum 90. A higher score represents increased severity and frequency of suicidal thoughts.
Suicide Attempts (SA) | Change from baseline to 6 months, 6 months to 9 months, and baseline to 9 months.
  Actual and interrupted suicide attempts (yes or no) using the Columbia-Suicide Severity Rating Scale (C-SSRS).
Suicidal Events (SE) | Change from baseline to 6 months, 6 months to 9 months, and baseline to 9 months.
  SE is defined as yes or no to any suicide attempt plus any ER visits due to suicidal ideation, and suicidal threats based on patient's own report and medical record, or by information gathered from the Child and Adolescent Services Assessment (CASA).
Depressive symptoms by self-report | Change from baseline to 6 months and baseline to 9 months.
  Level of depressive symptomatology using the Children Depression Inventory 2 (CDI-2). The CDI uses 27 items with a 4-point Likert type scale, the minimum score is 0 and the maximum 56. It evaluates symptoms such as depressive mood, hedonic capacity, vegetative sign, self-evaluation, and interpersonal behaviors. A higher score means higher level of depressive symptoms.
Depressive symptoms by clinical interview | Change from baseline to 6 months and baseline to 9 months.
  Depressive symptoms using the Children's Depression Rating Scale-Revised (CDRS-R). The CDRS-R is a 17-item interview assessment of depressive symptoms for school aged children and adolescents, with item rating between 1 (no difficulties) to 5 or 7 (clinically significant difficulties). The minimum raw score is 17 and the maximum 113. A higher score means higher level of depressive symptoms. It has been proposed that a score of ≥40 indicates depressive symptomatology comparable to a diagnosis of depression, whereas a score ≤28 was often used as indicative of remission within trials.

CONTACTS AND LOCATIONS:
Overall Officials: Yovanska Duarte-Velez, PhD, Principal Investigator — Brown University Health
Locations (1):
- Bradley Hasbro Children's Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Basic demographics and outcome measures will be uploaded to the NIMH Data Archive with a data dictionary.
Supporting Information: CSR
Time Frame: Data will be available starting 6 months after main study results publication.
Access Criteria: Researchers with access to the NIMH Data Archive will have access to the uploaded data. Data will also be made available to other researchers by request through a Data Sharing Agreement between institutions and as per NIH data sharing guidelines. The PI will also consult to anyone interested in replicating the intervention and study.

REFERENCES:
- [Background] Duarte-Velez Y, Torres-Davila P, Spirito A, Polanco N, Bernal G. Development of a treatment protocol for Puerto Rican adolescents with suicidal behaviors. Psychotherapy (Chic). 2016 Mar;53(1):45-56. doi: 10.1037/pst0000044. PMID 26928136
- [Background] Jimenez-Colon G, Duarte-Velez Y. Raising Children in Different Cultures: Working with Latinx Youth with Suicidal Behaviors and Their Families. R I Med J (2013). 2022 May 2;105(4):31-35. PMID 35476733
- [Background] Duarte-Velez Y, Jimenez-Colon G, Jones RN, Spirito A. Socio-Cognitive Behavioral Therapy for Latinx Adolescent with Suicidal Behaviors: A Pilot Randomized Trial. Child Psychiatry Hum Dev. 2024 Jun;55(3):754-767. doi: 10.1007/s10578-022-01439-z. Epub 2022 Oct 1. PMID 36183051